CLINICAL TRIAL: NCT03713892
Title: Phase I Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, PK, PD of CKD-504 in Single SAD and MAD in Healthy Korean and Caucasian Adult Male and Female Subjects
Brief Title: CKD-504 in SAD and MAD in Healthy Korean and Caucasian Adult Male and Female Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 175MAD17021
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — CKD-504; Histone Deacetylase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD-504 (Experimental): investigational Drug
  Interventions: Drug: CKD-504
- Placebo (Placebo Comparator): investigational Drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CKD-504 — orally administered once with investigational drug assigned on 1d morning with 240 mL of water
  Other Names: HDAC inhibitor
  Arms: CKD-504
Drug: Placebo — orally administered
  Arms: Placebo

SUMMARY:
To assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single and multiple ascending oral doses of CKD-504 compared to placebo in healthy Korean and Caucasian adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult Korean or Caucasian aged 19 to 45 (inclusive) years, at the time of screening.
* Subjects weighing ≥ 50 kg with BMI between 18 and 27 kg/m2 (inclusive) at screening visit.
* Subjects who agreed to voluntarily participate in this study and comply with all the protocol requirements by signing informed consent form after being informed of the nature of this study and understanding all aspects of this study.
* Subjects who were deemed as eligible subjects by investigators on their physical examination, laboratory findings, and medical examination by interview.

Exclusion Criteria:

* Subjects with a history of hypersensitivities to the drug, including investigational drugs or other drugs or with a history of clinically significant hypersensitivities.
* Subjects with a history of drug abuse or a positive urine screening for drug abuse.
* Subjects who have participated and taken investigational drug in any other clinical trial (including bioequivalence study) within three months prior to study drug administration.
* Subjects who have donated a unit of whole blood within 60 days or blood components within 30 days prior to study drug administration.
* Subjects judged ineligible for the study after a review of the clinical laboratory results by the investigator or for other reasons.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cmax of CKD-504 | Day1, Day2, Day3, Day4
  Peak Plasma Concentration (Cmax) of CKD-504
AUC of CKD-504 | Day1, Day2, Day3, Day4
  Area under the plasma concentration versus time curve (AUC) of CKD-504

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No